CLINICAL TRIAL: NCT00016432
Title: A Randomized Trial Evaluating The Effect Of Exemestane In Clinical Stage T1-3 N0-1 M0 Postmenopausal Breast Cancer Patients Completing At Least Five Years Of Tamoxifen Therapy
Brief Title: Exemestane in Treating Postmenopausal Women With Resected Stage I, Stage II, or Stage IIIA Breast Cancer Who Have Completed 5 Years of Tamoxifen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSABP B-33; CDR0000068640
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 1 (Experimental): Exemestane
  Interventions: Drug: exemestane
- Group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: exemestane — 25 mg for 5 years
  Arms: Group 1
Drug: Placebo — Placebo
  Arms: Group 2

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by reducing the production of estrogen by the tumor cells. It is not yet known whether exemestane is effective in preventing the recurrence of breast cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of exemestane in preventing cancer recurrence in postmenopausal women who have resected stage I, stage II, or stage IIIA breast cancer and have completed 5 years of tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the administration of 5 years of exemestane after 5 years of tamoxifen therapy is more effective than 5 years of prior tamoxifen therapy alone in prolonging disease-free survival, overall survival, and time to treatment failure in postmenopausal women with resected stage I, II, or IIIA breast cancer.
* Determine the effect of tamoxifen withdrawal on bone, in terms of height, fractures, and total alkaline phosphatase in these patients and on bone mineral density and bone biochemical markers in a subset of patients.
* Determine the effect of exemestane on bone loss after tamoxifen withdrawal in these patients.
* Evaluate the quality of life of a subset of these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral exemestane daily for 5 years.
* Arm II (closed as of 10/15/03): Patients receive an oral placebo daily for 5 years.

Quality of life is assessed at baseline and then every 6 months for 5.5 years.

Patients are followed every 6 months for 6 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 3,000 patients will be accrued for this study within 3 years and 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma of the breast at time of original diagnosis

  * Tumor confined to the breast and ipsilateral axilla on clinical exam (T1-3, N0-1, M0) (stage I-IIIA)
  * No ipsilateral lymph nodes clinically fixed to one another or to other structures (N2 disease) at time of original diagnosis
* Prior surgical resection, including 1 of the following:

  * Total mastectomy and axillary dissection (modified radical mastectomy) OR
  * Lumpectomy and axillary dissection

    * Prior post-lumpectomy breast radiotherapy required
  * Prior sentinel node biopsy allowed with the exception of the following:

    * If any sentinel node is histologically positive by hematoxylin and eosin (H & E) OR histologically suspicious on H & E and confirmed positive by immunohistochemistry then the patient must have a complete axillary dissection
  * Previously resected margins must be clear of invasive tumor and ductal carcinoma in situ
* Currently disease free
* Previously treated with tamoxifen for 57-66 months

  * Completed tamoxifen within the past 180 days
* No bilateral malignancy or mass in the opposite breast suspicious for malignancy unless biopsy proven negative
* No local, regional, or distant recurrence of disease or second primary breast malignancy (including contralateral breast cancer)
* No advanced disease at time of original diagnosis (e.g., ulceration, erythema, infiltration of the skin or underlying chest wall [complete fixation], peau d'orange, or skin edema of any magnitude)

  * Tethering or dimpling of the skin or nipple inversion allowed
* Current skeletal pain allowed if a bone scan and/or radiologic exam is negative for metastatic disease
* Hormone receptor status:

  * Primary tumor estrogen receptor (ER) positive AND/OR
  * Progesterone receptor positive
  * Borderline ER positive tumors allowed if previously treated with tamoxifen

PATIENT CHARACTERISTICS:

Age:

* Postmenopausal

Sex:

* Female

Menopausal status:

* Postmenopausal, defined as 1 of the following:

  * Prior bilateral oophorectomy
  * Absence of spontaneous menstrual cycle for more than 1 year
  * Follicle-stimulating hormone within the postmenopausal range if under 55 and had a prior hysterectomy without a bilateral oophorectomy

Performance status:

* Not specified

Life expectancy:

* At least 10 years

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin normal

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN
* Alkaline phosphatase less than 2 times ULN
* No systemic hepatic disease that would preclude study participation

Renal:

* Creatinine no greater than 1.5 times ULN
* No systemic renal disease that would preclude study participation

Cardiovascular:

* No systemic cardiovascular disease that would preclude study participation

Other:

* No other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, surgically treated carcinoma in situ of the cervix, or surgically treated lobular carcinoma in situ of the ipsilateral or contralateral breast
* No nonmalignant systemic disease that would preclude study participation
* No psychiatric or addictive disorder that would preclude informed consent
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior adjuvant chemotherapy allowed if administered concurrently with or prior to tamoxifen

Endocrine therapy:

* See Disease Characteristics
* No concurrent estrogen, progesterone, clomiphene, testosterone, gonadotropin-releasing hormone, oral contraceptives, selective estrogen-receptor modulators, or dehydroepiandrosterone (DHEA)

  * Estring or estrogen vaginal cream at 0.3 mg or 1/8 of an applicator applied vaginally 3 times a week allowed
* No other concurrent systemic hormonal therapy (e.g., tamoxifen or raloxifene)

Radiotherapy:

* See Disease Characteristics
* Prior post-mastectomy loco-regional radiotherapy or post-lumpectomy regional radiotherapy allowed

Surgery:

* See Disease Characteristics

Other:

* Prior participation in other adjuvant NSABP study allowed if study was reported in peer-review publication or tamoxifen was not a study drug
* Concurrent bisphosphonates or calcitonin for prevention or treatment of osteoporosis allowed
* Concurrent statins (simvastatin, pravastatin, fluvastatin, atorvastatin, or lovastatin) or other drugs to control lipid levels allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1598 (Actual)
Dates: Start 2001-05; Primary Completion 2003-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Every 12 months until breast cancer recurrence, second primary cancer or death from any cause.

SECONDARY OUTCOMES:
Overall survival | Death from any cause
Time to treatment failure | time from randomization to recurrence or contralateral second primary cancer
Bone measure as measured by total alkaline phosphatase, fracture history, and height measurement | measurements taken at regular intervals from randomization through 6 years following randomiztion

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (162):
- United States (150):
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Scripps Cancer Center, La Jolla, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute, Loma Linda, California
  - Pacific Shores Medical Group, Long Beach, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University Medical Center, Stanford, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Cancer Research Network Inc., Plantation, Florida
  - Oncology Hematology Consultants, Sarasota, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Center of Hawaii, Honolulu, Hawaii
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Illinois Oncology, Ltd., Belleville, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Norton Healthcare System, Louisville, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Staten Island University Hospital, Staten Island, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - Alamance Cancer Center, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center, Canton, Ohio
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - South Pointe Hospital - Cancer Care Center, Warrensville Heights, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Cancer Center, York, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Center for Oncology Research and Treatment, Medical City Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Camcare Health, Charleston, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (11):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Credit Valley Hospital, Mississauga, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
- MBCCOP - San Juan, San Juan, Puerto Rico

REFERENCES:
- [Result] Mamounas EP, Jeong JH, Wickerham DL, Smith RE, Ganz PA, Land SR, Eisen A, Fehrenbacher L, Farrar WB, Atkins JN, Pajon ER, Vogel VG, Kroener JF, Hutchins LF, Robidoux A, Hoehn JL, Ingle JN, Geyer CE Jr, Costantino JP, Wolmark N. Benefit from exemestane as extended adjuvant therapy after 5 years of adjuvant tamoxifen: intention-to-treat analysis of the National Surgical Adjuvant Breast And Bowel Project B-33 trial. J Clin Oncol. 2008 Apr 20;26(12):1965-71. doi: 10.1200/JCO.2007.14.0228. Epub 2008 Mar 10. PMID 18332472
- [Result] Mamounas E, Jeong J-H, Wickerham L, et al.: Benefit from exemestane (EXE) as extended adjuvant therapy after 5 years of tamoxifen (TAM): intent-to-treat analysis of NSABP B-33. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-49, S22, 2006.